CLINICAL TRIAL: NCT00055705
Title: A Phase I Clinical Trial To Assess The Safety And Efficacy Of Intraperitoneal PV701 Administrations In Patients With Advanced Or Recurrent Malignancy Largely Confined To The Peritoneal Cavity
Brief Title: PV701 in Treating Patients With Advanced or Recurrent Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000270801; MSKCC-02080; NCI-1617
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2004-08

CONDITIONS: Cancer
Keywords: recurrent ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer; recurrent colon cancer; stage IV colon cancer; ovarian sarcoma; recurrent ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent endometrial carcinoma; stage IV endometrial carcinoma; recurrent uterine sarcoma; stage IV uterine sarcoma; ovarian stromal cancer; recurrent rectal cancer; stage IV rectal cancer; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; gastrointestinal stromal tumor; advanced malignant mesothelioma; recurrent malignant mesothelioma; recurrent gastric cancer; stage IV gastric cancer; carcinoma of the appendix; small intestine adenocarcinoma; small intestine leiomyosarcoma; small intestine lymphoma; recurrent small intestine cancer; recurrent gallbladder cancer; unresectable gallbladder cancer; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Colonic Neoplasms; Endometrial Neoplasms; Rectal Neoplasms; Gastrointestinal Stromal Tumors; Mesothelioma, Malignant; Stomach Neoplasms; Appendiceal Neoplasms; Gallbladder Neoplasms; Carcinoma, Hepatocellular

INTERVENTIONS:
Biological: PV701

SUMMARY:
RATIONALE: PV701 may be able to kill tumor cells while leaving normal cells undamaged.

PURPOSE: Phase I trial to study the effectiveness of PV701 in treating patients who have advanced or recurrent ovarian epithelial, fallopian tube, primary peritoneal, colorectal, or other cancer found primarily within the peritoneal cavity.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose-limiting toxicity and maximum tolerated dose of intraperitoneal PV701 after desensitization in patients with advanced or recurrent malignancy largely confined to the peritoneal cavity these patients.
* Determine the optimal desensitization dose of intravenous PV701 in these patients.
* Determine the safety of this drug, in terms of cumulative toxicity, in these patients.
* Determine, preliminarily, the antitumor activity of this drug in these patients.
* Determine the presence and duration of viral shedding, viremia, and immunogenicity of this drug.

OUTLINE: This is an open-label, dose-escalation study comprising 2 different treatment schedules.

* Schedule I (optimal desensitization dose): Patients receive PV701 IV over 30 minutes on day 1 followed by intraperitoneal (IP) PV701 on days 4, 7, and 9. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of PV701 IV and IP until the optimal desensitization dose (ODD) is determined. The ODD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity (DLT).

* Schedule II (maximum tolerated dose):Patients receive the same regimen as in schedule I using PV701 IV at the ODD.

Cohorts of 3-6 patients receive escalating doses of PV701 IP until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience DLT.

PROJECTED ACCRUAL: A total of 3-50 patients will be accrued for this study within 10-17 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histological confirmation of 1 of the following:

  * Ovarian epithelial carcinoma
  * Fallopian tube cancer
  * Primary peritoneal cancer
  * Advanced colorectal carcinoma
  * Other malignancy confined to the peritoneal cavity or peritoneal surfaces
* No lesion greater than 2 cm in greatest diameter based on surgical re-assessment
* Low burden of tumor in the abdominal or pelvic cavities and no clinically significant ascites
* Received potentially effective therapy when available (e.g., platinum/taxane for ovarian cancer, fluoropyrimidine-based therapy for colorectal cancer)
* No concurrent hematological malignancy (e.g., chronic lymphocytic leukemia or non-Hodgkin's lymphoma)
* No bilateral adrenal metastases
* No adrenal metastases in the remaining adrenal gland after adrenalectomy (including radical nephrectomy)
* No lung tumors 5 cm or more
* No pleural effusions (at least 25% of hemithorax) by radiography
* No CNS metastases by CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 9 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 1.5 times ULN
* No uncontrolled hepatic dysfunction
* No active hepatitis B or C

Renal

* See Disease Characteristics
* Creatinine no greater than 1.6 mg/dL AND/OR
* Creatinine clearance at least 50 mL/min
* No uncontrolled renal dysfunction

Cardiovascular

* No uncontrolled cardiovascular dysfunction
* No myocardial infarction within the past 6 months
* No life-threatening arrhythmias within the past 6 months

Pulmonary

* See Disease Characteristics
* No uncontrolled pulmonary dysfunction
* No pulmonary atelectasis (lobar)
* No pulmonary infiltrates (lobar)
* No pulmonary consolidation (lobar or segmental)
* No baseline grade II dyspnea

Adrenal

* See Disease Characteristics
* No uncontrolled adrenal dysfunction
* No known adrenal insufficiency

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled gastrointestinal dysfunction
* No neurological dysfunction
* No serious medical or psychological condition that would preclude study participation or increase the risk of adverse effects of the study treatment
* No history of serious immunodeficiency
* No active uncontrolled bacterial infection (including asymptomatic urinary tract infection)
* No contraindication to intraperitoneal therapy including the following:

  * Intra-abdominal infection
  * Dense widespread adhesions
  * Peritonitis
  * Periumbilical infection
  * Bowel obstruction
  * Ileostomy
* No hypersensitivity to eggs
* No continued contact with live birds (e.g., poultry farmers, veterinarians, laboratory technicians, pet store owners, breeders)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No more than 3 prior cytotoxic chemotherapy regimens
* More than 30 days since prior chemotherapy

Endocrine therapy

* More than 14 days since prior systemic corticosteroids

Radiotherapy

* More than 30 days since prior radiotherapy

Surgery

* See Disease Characteristics
* No prior complete or partial lobectomy with removal of lung tissue at least segmental size
* No prior organ allograft

Other

* Recovered from prior therapy
* More than 14 days since prior antiviral medication
* More than 4 weeks since prior immunosuppressive drugs
* No other concurrent investigational drugs
* No concurrent chronic immunosuppressive drugs (e.g., cyclosporine)
* No vaccination for influenza within 48 hours of study drug administration
* No concurrent hypoglycemic agents
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-01

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spriggs, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States